CLINICAL TRIAL: NCT04412200
Title: Randomized Controlled Study to Evaluate the Effect of Hyperbaric Oxygen Therapy (HBOT) on Treg-CD4+Cells, Cytokines Profile, and Beta Cells Reserve in New-onset Type-1 Diabetes Mellitus
Brief Title: Efficacy of Hyperbaric Oxygen Therapy (HBOT) in New-onset Type-1 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0290-19-ASF
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: T1DM
Keywords: Hyperbaric chamber; autoimmune disease; inflammation; recent onset autoimmune diabetes; beta cells; diabetes mellitus type 1; pediatrics
MeSH Terms: conditions — Autoimmune Diseases; Inflammation; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric oxygen chamber Arm (Experimental): Patients will be randomized at a ratio of 2:1, to hyperbaric chamber (100% oxygen at 2 ATA)
  Interventions: Device: Hyperbaric oxygen chamber (HBOC)
- Control arm (No Intervention): control group will receive common practice management.

INTERVENTIONS:
Device: Hyperbaric oxygen chamber (HBOC) — HBOC group will receive 100% oxygen at 2 ATA for 90 min with 5 min air breaks every 20 min at each session. Intensive management period includes 60 daily sessions, 5 days per week within 12 weeks,
  Arms: Hyperbaric oxygen chamber Arm

SUMMARY:
Type 1 Diabetes Mellitus (T1DM) is caused by an autoimmune process that progressively destroys the pancreatic β-cells, and leads to dependence on multiple daily insulin subcutaneous injections according to glucose measurements and dietary restrictions, leading to short and long term complications. Current data demonstrate that even modest preservation of β-cell function and endogenous production of insulin (marked by C-peptide) may result in meaningful clinical benefits including lower rates of complications, improved metabolic control, reduced insulin injections, and improved quality of life.

Objective:

1. To assess the effect of HBOT on Treg, mesanchymal stem cells, and pro-inflammatory cytokines ratio in pediatric population with new-onset T1DM Secondary
2. To assess the effect of HBOT on beta cell reserve in pediatric population with new-onset T1DM
3. To assess the effect of HBOT on glycemic control parameters including time in range, HbA1c and daily insulin dose, in the pediatric population with new-onset T1DM

Study design:

Randomized, controlled study of pediatric and young adults patients who have been newly diagnosed with type 1 diabetes within 12 weeks prior to randomization (4-6 weeks from screening) and express peak C-peptide ≥ 0.2 pmol/ml Subjects will be randomized to hyperbaric oxygen chamber (HBOC) group and to a non-intervention, control group. Both groups will be managed similarly by carbohydrate counting and basal bolus insulin administration, based on their interstitial glucose levels by glucose continuous glucose monitoring system (CGMS) and carbohydrate counting before meals.

The intervention protocol includes 12 weeks of intensive management, and 12 weeks of follow up.

During the intensive management period - for 12 weeks, the HBOC group will receive 100% oxygen at 2 ATA for 90 min with 5 min air breaks every 20 min at each session. Intensive management period includes 60 daily sessions, 5 days per week within 12 weeks, During the intensive management period - for 12 weeks, the control group will receive common practice managemnt.

All will be instructed to inject insulin pre-meals according to carbs-counting, and CGMS. Insulin will be administered by subcutaneous continuous insulin infusion (SCII) or by pens with CLIPSULIN only, for accurate daily dose of insulin recording.

Along the 24 weeks of the study several parameters will be assessed at pre-defined time points .

1. Immune system parameters will be assessed by blood levels of T-regulatory cells, diabetes auto-antibody and inflammatory cytokines.
2. Pancreatic β cells function will be evaluated by measurements of blood area under the curve (AUC) C-peptide, peak C-peptide, and basal proinsulin/c-peptide ratio.
3. glycemic control parameters will be evaluated by CGMS data regarding time spent in glycemic range, hypoglycemic and hyperglycemic ranges, total daily dose of insulin according to CLIPSULIN , and blood tests for glycated hemoglobin (HbA1c).
4. Microbiome changes will be assessed by stool samples.

Expected significance: the study suggests a safe modality used clinically among adults and other paediatric conditions, for the possible solution of an unmet urgent medical need, studied successfully in an animal model. The study is designed to be powered to answer the question of efficacy, and in addition, addresses the mechanisms by which it may halt the progression of β cell destruction in new onset T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian willing and able to sign an informed consent
* Participant willing and able to sign an assent
* Diagnosed with type 1 diabetes within 12 weeks prior to randomization
* Treated with insulin by basal-bolus regimen (injections or pump)
* Peak C-peptide ≥ 0.2 pmol/ml
* At least 1 positive diabetes auto-antibody
* No significant abnormalities in hematology and serum chemistry according to the investigator's judgment, taking into consideration the potential effects of the diabetic illness
* No significant abnormalities in urinalysis, taking into considerations the potential effects of the diabetic illness
* For females of child bearing potential: whose screening pregnancy test is negative and who are using contraceptive methods deemed reliable by the investigator

Exclusion Criteria:

* Planned major surgery within the study period
* Clinically significant inter-current illnesses, including (but not limited to): lung, cardiac, hepatic, renal, eye, neurological, hematological, neoplastic, immunological, skeletal or other, that in the opinion of the investigator, could interfere with the safety, compliance or other aspects of this study. Patients with well-controlled, chronic diseases could be possibly included after consultation with the investigator at site.
* Presence of psychiatric/ mental disorder or any other medical disorder which might impair the patient's ability to give informed consent or to comply with the requirements of the study protocol
* Participation in another interventional clinical trial
* Inability to attend scheduled clinic visits and/or comply with the study protocol
* Current use of any medication known to influence glucose tolerance (e.g., β-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine anti-malarial drugs, lithium, niacin, metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors or amylin).
* Lung disease, middle ear disease, inner ear disease, history of epileptic seizures or any other condition that based on the physician clinical judgment is not suitable to get the hyperbaric treatment.
* Any other factor that, in the opinion of the investigator, would prevent the patient form complying with the requirements of the protocol.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Regulatory T cells and B cells | 24 weeks
Cytokine secretion | 24 weeks
  by stimulated peripheral blood mononuclear cells cultured with LPS or PHA for 72 hours, and in supernatant will be measured by relevant commercial ELISA kits

SECONDARY OUTCOMES:
insulin daily dose (IDD) unit/kg/d | 24 weeks
  Difference between groups in achievement of glycemic targets according to ITDD, with a lower ITDD. assessed by: mean and SD of glucose, CV, time spent in range >70%, and time spent at hypoglycemic range < 1% at end of treatment periods, IDD according to weight.
C-max of stimulated C peptide | 24 weeks
  Difference between treatment groups (HBOT/SHBC) in change of β cell function (measured by C-max of stimulated C peptide) from screening to end of study (24 weeks).
AUC of stimulated C peptide | 24 weeks
  Difference between treatment groups (HBOT/SHBC) in change of β cell function (measured by AUC of stimulated C peptide) from screening to end of study (24 weeks).

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Asaf harofe medical center, Tzrifin
  - Assaf Haroffeh Medical center, Zrifin